CLINICAL TRIAL: NCT05441631
Title: Dysglycemia and COVID-19 Disease: A Reciprocal Relationship. Can Intensive Insulin Therapy Cut This Vicious Circle?
Brief Title: Can Intensive Insulin Therapy Improve Outcomes of COVID-19 Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amr M. El Hammady, Assistant professor of Internal Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 1.6.2020
Record Dates: First submitted 2022-06-18; First posted 2022-07-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Dysglycemia
MeSH Terms: conditions — COVID-19 | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intensive insulin therapy (Active Comparator)
  Interventions: Drug: Insulin
- Conventional insulin therapy (Active Comparator)
  Interventions: Drug: Subcutaneous Insulin

INTERVENTIONS:
Drug: Insulin — * Preparation: 50 IU of rapidly acting insulin in 50 ml of 0.9% saline solution was delivered through a 50-ml syringe-driven pump.
  * Monitoring: The insulin dose was adjusted to whole-blood glucose levels using glucometer every hour and insulin infusion was continued till BG level (Targeted level) was 80-110 mg, and then BG levels were estimated four-hourly
  * Insulin dose was titrated according to the Leuven titration protocol (15)
  Arms: Intensive insulin therapy
Drug: Subcutaneous Insulin — * Insulin dose was titrated according to the Blood glucose level
  * monitoring according to glucose in urine
  Arms: Conventional insulin therapy

SUMMARY:
Evaluation of the reciprocal relation between hyperglycemia/diabetes mellitus (HG/DM) and COVID-19 disease and the effect of mode of insulin therapy; intensive (IIT) or conventional (CIT) on patients' outcomes All patients admitted to the quarantine hospitals with mild-severe COVID disease were evaluated using the COVID-GRAM Critical Illness Risk Score and gave blood samples for estimation of random blood glucose. Diabetic patients and non-diabetic patients with persistent HG were randomly divided according to mode of IT. Patients who were free HG were included as control normoglycemic (NG) patients. Study outcomes included the incidence of progress to critical illness and mortality rate (MR), and the effect of IT on such outcomes

DETAILED DESCRIPTION:
All patients admitted to the quarantine department at Benha University hospital and quarantine hospitals all over the Qalyubia Governorate were eligible for evaluation for exclusion criteria. Taking on the precautions according to the instruction of the Ministry of Health on dealing with suspected or confirmed COVID patients and with the application of conditions of Infection Control Programs and considering the personal protective equipment, clinical, radiological, and laboratory evaluation were undertaken.

1. COVID-19 disease severity grading Patients were categorized according to the guidelines of the National Institutes of Health (NIH) and patients with pre-symptomatic infection or critical disease severity were excluded, while patients with mild-to-severe disease severity grade were enrolled in the study: Mild disease was defined as the presence of any of the signs and symptoms of COVID-19 without shortness of breath, dyspnea, or abnormal chest imaging. The moderate disease was determined by the presence of evidence of lower respiratory disease during clinical assessment or imaging, but oxygen saturation (SpO2) was ≥94% on room air at sea level. Patients were diagnosed as having the severe disease if SpO2 was <94% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, respiratory frequency >30 breaths/min, or lung infiltrates >50% (10).
2. Diagnosis of hyperglycemia Stress hyperglycemia was defined according to the American Association of Clinical Endocrinologists and American Diabetes Association Consensus Statement on Inpatient Glycemic Control, as transient BG level at the time of admission >140 mg/dl that subsided on relief of stress and apprehension, but if BG persisted >140 mg/dl at 6-hr after admission it is persistent hyperglycemia and needs intervention (11). For diagnosis of hyperglycemia and determination of baseline BG level of diabetic patients blood samples were obtained at admission and 6-hr thereafter for non-diabetic and put in a tube containing sodium fluoride (2 mg sodium fluoride/ ml blood) to prevent glycolysis till estimation of BG levels using glucose oxidase method (12).
3. COVID-GRAM Critical Illness Risk Score At the time of admission, the risk for progression to critical COVID-19 illness was evaluated by one of the authors and the determined risk remained uncovered till the end of the study for comparative purposes. The risk of progression to critical illness depended on the three outcomes defined by Liang et al. (13) as admission to the ICU, need for invasive mechanical ventilation (IMV), or death. The risk of progression to critical illness was determined qualitatively as low, medium, or high and quantitatively as risk percentage using the COVID-GRAM Critical Illness Risk (CG-CIR) Score that can be computed depending on clinical, radiological, and laboratory findings at the time of admission using an online calculator (14).

Patients' grouping

* Diabetic group: includes patients with definite DM and maintained on anti-diabetic therapy, either oral hypoglycemic or insulin therapy. Patients were divided according to the type of DM as T1D or T2D groups.
* Non-diabetic group: included patients who denied any history of DM or receiving antidiabetic therapy and were categorized as normoglycemic (NG) if their at admission random BG was <140 mg/dl or had stress hyperglycemia that disappeared at the 6-hr estimation of BG (NG Group), and hyperglycemic if their at admission BG level was >140 mg/dl and persisted at 6-hr estimation (HG Group).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic
* Non-diabetic
* Confirmed COVID-19 disease both by PCR diagnosis of viral RNA and by CT diagnosis of COVID- associated pneumonia.

Exclusion Criteria:

* Patients younger than 18 years,
* Patients admitted with critical illness requiring immediate admission to ICU,
* Patients deceased before evaluation,
* Patients who had autoimmune diseases or were maintained on immunosuppressive therapy,
* Patients with chronic medical diseases other than DM,
* Patients requiring surgical interference for emergency conditions, and
* Patients who had cancer or were maintained anticancer therapy were excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The relation between application intensive insulin therapy and patients' survival | 12 months
  The relation between intensive insulin therapy and patients outcome regarding deuteration to Critical illness grade and mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, El- Qalyobia, Egypt

IPD SHARING:
Plan to Share IPD: No